CLINICAL TRIAL: NCT01041846
Title: A Prospective Multicenter Observational Study for Dacogen Treatment in Patients With Myelodysplastic Syndrome
Brief Title: A Study for Dacogen Treatment in Patients With Myelodysplastic Syndrome
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015895; DECKOR5002 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2009-12-17; First posted 2010-01-01 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; Dacogen; Decitabine; Epigenetic therapy; Hypomethylating agent
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Decitabine
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Patients receiving 20 mg/m2 of decitabine injection intravenously (into a vein) once daily for 5 days every 4 weeks will be observed.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of decitabine (Dacogen) intravenous injection in patients with Myelodysplastic Syndrome.

DETAILED DESCRIPTION:
This is a prospective (in which the patients are first identified and then followed forward as time passes), multi-center (study conducted at multiple sites), observational study (a scientific study to make a clear and easy understanding of the cause and effect relationship) to evaluate the effectiveness and safety information of a 5 day decitabine (Dacogen) regimen in patients with Myelodysplastic Syndrome. This study consist of 3 phases; pre-treatment phase, treatment phase and end of treatment (Day 28~61 after last administration of Dacogen). The patients will receive decitabine intravenous injection 20 mg/m2 one hour once daily for 5 consecutive days for every 4 weeks. Safety evaluations including adverse events and clinical laboratory tests and will be evaluated with adverse events reported for the period ranging from informed consent and during the study to the end of treatment visit including 56 days (8 weeks) after the last administration of the clinical study treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with (primary or secondary) Myelodysplastic Syndrome including chronic myelomonocytic leukemia (CMML) with an International Prognostic Scoring System more than or equal to Interferon-1

* Patients who have never treated with hypomethylating agent (azacitidine and decitabine)
* Female patients who are postmenopausal or received contraceptive operation or refrain from sexual relations.
* Women of childbearing potential should conduct an effective method of birth control as defined in protocol, in case of male patients who will not have a baby within 2 months after the completion of decitabine therapy

Exclusion Criteria:

* Patients diagnosed with acute myelogenous leukemia (bone marrow stem cell counts exceeding 20 %) or other progressive malignant diseases
* Patients with active infection of virus or bacteria
* Patients who used to be treated with azacitidine or decitabine
* Patients who are hypersensitive to excipients of decitabine
* Patients who are pregnant and breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who signed the subject informed consent form among the patients with myelodysplastic syndrome who were treated with decitabine
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete remission | Up to 61 days
  The complete response includes the evaluations of Bone marrow aspiration and biopsy (less than or equal to 5 percents myeloblast), persistent dysplasia and peripheral blood.
Number of patients with partial remission | Up to 61 days
  The partial response includes all complete remission evaluating parameters with the exception of bone marrow blasts are decreased by more than or equal to 50 percents over pretreatment but still more than 5 percents and cellularity (the state of a tissue or other mass as regards the number of its constituent cells) and morphology (examination of structure)
Number of patients with hematological improvement | Up to 61 days
Response rate | After 4 cycles and end of treatment
  Response rate is the combination of complete remission, partial remission and hematological improvement and performed according to the response criteria of 'International Working Group 2006' which is standardized criteria for assessing response are essential to ensure comparability among clinical trials for patients with MDS.

SECONDARY OUTCOMES:
Cytogenetic response rate | Up to 61 days
Overall survival rate | Up to 61 days
  Overall survival will be evaluated from the registration day to death.
Time to acute myeloid leukemia evolution | Up to 61 days
  The time of progression from myelodysplastic syndromes to acute myeloid leukemia.
Number of patients with progression-free survival status | Up to 61 days
  Hospitalization or undergoes surgical procedure due to disease progression.
Number of patients with adverse event | Up to 61 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

REFERENCES:
- [Derived] Jung KS, Kim YJ, Kim YK, Park SK, Kim HG, Kim SJ, Park J, Choi CW, Do YR, Kim I, Park S, Mun YC, Jeong SH, Kim MK, Yi HG, Chang MH, Kim SY, Lee JH, Jang JH. Clinical Outcomes of Decitabine Treatment for Patients With Lower-Risk Myelodysplastic Syndrome on the Basis of the International Prognostic Scoring System. Clin Lymphoma Myeloma Leuk. 2019 Oct;19(10):656-664. doi: 10.1016/j.clml.2019.06.003. Epub 2019 Jun 27. PMID 31375393
- [Derived] Lee JH, Jang JH, Park J, Park S, Joo YD, Kim YK, Kim HG, Choi CW, Kim SH, Park SK, Park E, Min YH. A prospective multicenter observational study of decitabine treatment in Korean patients with myelodysplastic syndrome. Haematologica. 2011 Oct;96(10):1441-7. doi: 10.3324/haematol.2011.046078. Epub 2011 Jun 9. PMID 21659363
- See also: A Prospective, Multicenter, Observational Study of Dacogen Treatment in Patients with Myelodysplastic Syndrome — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=337&filename=CR015895_CSR.pdf